CLINICAL TRIAL: NCT04163068
Title: The Improving Cancer Aftercare Study. Using Patient and Caregiver Experiences to Assess Treatment Burden and Inform Health Service Design for People After Prostate and Colorectal Cancer. A Qualitative Semi-structured Interview Study.
Brief Title: The Improving Cancer Aftercare Study.
Acronym: ICAS
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-078-19
Record Dates: First submitted 2019-11-04; First posted 2019-11-14 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Prostate Cancer
Keywords: cancer; survivorship; qualitative interviews; treatment burden; cancer aftercare; self management
MeSH Terms: conditions — Colorectal Neoplasms; Prostatic Neoplasms; Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview with researcher: All participants will participate in an interview with a researcher
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — The interview will last approximately 45 minutes, will be audio-recorded, transcribed, and analysed

SUMMARY:
This is a qualitative interview study that aims to understand treatment burden in individuals who have experienced prostate or colorectal cancer treatment within the past five years. We intend to use patient and caregiver experiences to co-design interventions to optimise cancer aftercare.

Treatment burden is the workload of healthcare for patients and the consequences of this workload on patient function. Treatment burden has been associated with negative outcomes in stroke, heart failure, diabetes, and renal failure. Cancer is increasingly becoming a chronic condition, and involves a variety of self-management tasks for patients and their caregivers. In this study investigators will investigate treatment burden in people after prostate and colorectal cancer. Investigators will seek to understand patient and caregiver perceptions about cancer aftercare, and ways that services could be redesigned and improved to reduce treatment burden, and improve patient outcomes.

We will undertake a qualitative interview study, recruiting patients from general practices and oncology outpatient clinics who have completed potentially curative treatment for prostate or colorectal cancer, or who are on active surveillance or hormonal therapies for localised or locally advanced prostate cancer. We will purposively sample, to ensure that participants with comorbidities, those from lower socioeconomic groups, and rural dwellers are adequately represented. We will conduct interviews according to a schedule, informed by conceptual models of burden of treatment, Schwarzer's Health Action Process Approach, and Normalisation Process Theory.

Interviews will be filmed and/or audio-recorded and transcribed. Framework and thematic analysis will be used to analyse and synthesise the data. Participants will be given the chance to comment on outputs and findings (triangulation).

Investigators plan to use the results of this study, and excerpts from video interviews during co-design events, and to create new interventions to optimise aftercare for patients with prostate and colorectal cancer.

DETAILED DESCRIPTION:
The number of individuals surviving for more than five years following a cancer diagnosis is steadily rising. Cancer is often a long-term condition. Individuals living beyond a cancer diagnosis are required to participate in a range of self-management activities, including (and not limited to) managing symptoms and comorbidities, self-monitoring for recurrence, adjusting to life beyond cancer/managing psychological sequelae, taking medications, attending follow-up appointments, and addressing unhealthy behaviours.

Treatment burden is the workload of healthcare for patients, and the effect that this work has on patient functioning and well-being. In the 1960s, Thomas Creer recognised that patient participation in their own healthcare was important in achieving disease control in paediatric asthma. Since then, "self-management" has been extensively researched and conceptualised. In the 1980s, Corbin and Strauss characterised three strands of "work" for people with chronic conditions: medical management, for example adhering to medication regimens and attending appointments; behavioural management, such as adopting healthier lifestyle practices; and the emotional management of adapting to a long-term condition.

Increasing patient participation in self-management has mostly been viewed as a positive strategy through which to improve health outcomes, reduce medical paternalism, and delegate some tasks away from over-burdened health and social care systems. Treatment burden is a relatively recent concept which highlights the potentially deleterious effects of increasing patient workload. Treatment burden is becoming increasingly relevant as more people survive into old age, often with combinations of comorbidities (including cancer) for which there are multiple available therapeutic agents and complex self-management regimens.

In diabetes, renal failure, heart failure, and stroke, there is increasing evidence that increased treatment burden is associated with reduced quality of life, non-adherence to therapeutic regimes, and wasted resources. Treatment burden is modified by patient capacity: those with lower self-efficacy, low levels of social support, financial difficulties, and competing personal workload can experience increased treatment burden. In cancer, certain large and distinct demographic groups, particularly rural dwellers and the socially deprived, have poorer survival after a cancer diagnosis. The mechanisms of these inequities have not been adequately explained.

It is feasible that treatment burden could modify interactions with health services, engagement with survivorship activities, and ultimately, cancer outcomes.

Treatment burden is a relatively recent concept which is under-explored in in cancer survivors.

The objectives of this study are:

1. To investigate patient perceptions of treatment burden after prostate and colorectal cancer.
2. To determine sources of treatment burden in prostate and colorectal cancer survivors, their interactions, and the perceived consequences of treatment burden.
3. To utilise key concepts from the interviews to build a video narrative, featuring video excerpts from participants to ensure that their voices reach a wider audience, including professionals. We will use these narratives to improve cancer services through co-design.

Qualitative interview will be conducted with approximately 40 patients, with or without linked caregivers. They will be transcribed verbatim, and analysed using Framework and thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have a history of prostate or colorectal cancer within the past five years (we are interested in recent experiences and most individuals with colorectal cancer are discharged by five years from hospital follow up)
* Individuals who have or have had localised or locally advanced disease, treated by any method, including and not limited to active surveillance, surgery, radiotherapy, or chemotherapy.
* Adult age 18 years or over
* Caregivers for an individual who meets the above criteria, who are aged 18 years or over.

Exclusion Criteria:

* • Individuals who do not wish to participate

  * Individuals who do not understand and/or speak English
  * Individuals with significant cognitive impairment, learning difficulty, or communication difficulty such that understanding the nature of the study, the interview questions, or participating in an interview would not be practical
  * Presence of distant metastases at the time of recruitment, which are being treated with palliative intent (treatment and follow up for these individuals has different aims and format)
  * Individuals who are currently undergoing or on waiting lists for chemotherapy, radiotherapy, or surgery (for their colorectal or prostate cancer)
  * Caregivers who do not have a linked patient participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors of prostate or colorectal cancer and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Treatment burden | 12 months
  Patient and caregiver perceptions of treatment burden assessed through semi-structured interviews and analysed by Framework and thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Adam, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adam R, Duncan L, Maclennan SJ, Locock L. Treatment burden in survivors of prostate and colorectal cancers: a qualitative interview study. BMJ Open. 2023 Mar 3;13(3):e068997. doi: 10.1136/bmjopen-2022-068997. PMID 36868591